CLINICAL TRIAL: NCT05837416
Title: Comparative Study of the Effect of Oxidant Gel and Anti-oxidant Gel on Wound Healing After Gingival Depigmentation. (A Randomized Controlled Clinical Trial)
Brief Title: Effect of Oxidant Gel and Anti-oxidant Gel on Wound Healing After Gingival Depigmentation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Metwally Shafik Metwally, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16223
Record Dates: First submitted 2023-04-15; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Gingival Pigmentation
Keywords: Oxidant Gel; Anti-oxidant Gel; Gingival depigmentation
MeSH Terms: interventions — Coe-Pak

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor and biostatistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxygen Releasing Oral Gel (blue®m) with Coe-Pak dressing (Experimental): topical application of Oxygen Releasing Oral Gel (blue®m) on the surgical site followed by Coe-Pak immediately after gingival depigmentation surgery, then 1 week postoperatively
  Interventions: Drug: blue®m Gel
- Nano-emulsion complex propolis and vitamin C (NBF GINGIVAL GEL®) with Coe-Pak dressing (Experimental): topical application of Nano-emulsion complex propolis and vitamin C (NBF GINGIVAL GEL®) on surgical site followed by Coe-Pak immediately after surgery, then 1 week postoperatively
  Interventions: Drug: NBF GINGIVAL GEL®
- COE-PAK periodontal dressing only (Active Comparator): Periodontal dressing (COE-PAK) will be applied on surgical site only .
  Interventions: Drug: COE-PAK™

INTERVENTIONS:
Drug: blue®m Gel — Oxygen will be released after application Oxygen Releasing Oral Gel (blue®m gel) creating a partially high oxygen pressure (pO2), which aids in restoring the micro-environment for a healthy oral cavity
  Other Names: Oxygen Releasing Oral Gel
  Arms: Oxygen Releasing Oral Gel (blue®m) with Coe-Pak dressing
Drug: NBF GINGIVAL GEL® — Anti-oxidant gel (Nano-emulsion complex propolis and vitamin C - NBF GINGIVAL GEL®) is a nano bio fusion gel containing propolis, nano vitamin C, E and herb extract
  Other Names: nano bio fusion gingival gel
  Arms: Nano-emulsion complex propolis and vitamin C (NBF GINGIVAL GEL®) with Coe-Pak dressing
Drug: COE-PAK™ — It is non eugenol periodontal dressing. It is supplied in two tubes, the contents of which are mixed immediately before use. One tube contains zinc oxide, oil, a gum, and lorothidol. The other tube contains liquid coconut fatty acids thickened with colophony resin and chlorothymol
  Arms: COE-PAK periodontal dressing only

SUMMARY:
To evaluate effect of Oxidant (Oxygen Releasing Oral Gel) with Coe-Pak versus Anti-oxidant (Nano-emulsion complex propolis and vitamin C gel) with Coe-Pak on wound healing, pain, patient satisfaction after gingival depigmentation

DETAILED DESCRIPTION:
Gingival depigmentation is considered a periodontal plastic surgery, in which gingival hyperpigmentation is eliminated. The scalpel surgical method is one of the most cost-effective methods, easiest and does not need broad equipment. However, scalpel surgery leads to bleeding during and after surgery, and the surgical area has to be covered with periodontal dressing for 7-10 days. Periodontal dressings are used around the necks of the teeth and surrounding tissue to cover the wound. Non-eugenol dressings are now the most commonly used periodontal dressings include Coe-Pak, Cross Pack, Peripac, Septopack, PerioCare, Perio Putty and Periogenix. Anti-oxidant gel (Nano-emulsion complex propolis and vitamin C - NBF GINGIVAL GEL®) is a high efficiency nano bio fusion gel containing propolis, nano vitamin C, E and herb extract. Anti-oxidant power of nano Vitamin C (NBF GINGIVAL GEL®) is ten times more effective in hundred times smaller amounts, than Vitamin C by itself. Vitamin C collaboratives with Vitamin E and preserves cell membranes integrity. Propolis has antioxidant effect due to its radical scavenging ability, which was more efficient than antioxidant effect of vitamin C. it also enhances synthesis of collagen due to the presence of iron and zinc elements. it has proven to increase healing of epithelial tissues. The presence of oxygen in Oxygen Releasing Oral Gel (blue®m gel) enhances cellular metabolism, collagen synthesis, antibacterial activity, angiogenesis, revascularization, and the release of growth factors, it also helps keratinized tissue formation and has antimicrobial effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with anterior maxillary or mandibular physiologic gingival pigmentation
* Systemically healthy patients
* Good oral hygiene, Plaque index less than 15%.
* Cooperative patients able and accept to come for follow up appointments

Exclusion Criteria:

* Any interim intervention that may have affected any of the outcomes of interest.
* Pregnant and lactating females.
* Smokers
* Patients reporting systemic conditions that may cause hyperpigmentation (eg.Addison's disease) or on medications (eg. Corticosteroids)
* Patients reporting systemic conditions that may compromise healing (eg. Diabetes)
* Patients with poor oral hygiene.
* Any known allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
wound healing | Change in healing from baseline up to 4 weeks
  Assessment of healing using the healing index scale by Landry with scale starting from (1 for very poor healing and 5 excellent healing).Postoperatively clinical photographs will be taken.

SECONDARY OUTCOMES:
Post-operative Pain Assessment | 7 days
  pain score will be measured at 1st week . Visual Analogue Scale (VAS) will be used to evaluate pain with score starting from 0 (minimal pain ) to 10 ( maximum pain). Questionnaire
Post-operative Pain Assessment | 14 days
  pain score will be measured at 2nd week. Visual Analogue Scale (VAS) will be used to evaluate pain with score starting from 0 (minimal pain ) to 10 ( maximum pain) . Questionnaire
Patient Satisfaction | 30 days
  Questionnaire (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Darhous, PHD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No